CLINICAL TRIAL: NCT03583840
Title: Effectiveness of a Web-based Intervention to Promote Health Screening in Men: A Community-based Randomised Controlled Trial
Brief Title: Effectiveness of a Web-based Intervention to Promote Health Screening in Men
Acronym: ScreenMen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Malaya (Other)
Collaborators: Leeds Beckett University (Other); University of Sheffield (Other); The University of New South Wales (Other)
Responsible Party: Principal Investigator, Professor Ng Chirk Jenn, Professor Dr, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RP041A-15HTM
Record Dates: First submitted 2018-06-18; First posted 2018-07-11 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Mass Screening; Preventive Health Services
Keywords: men's health; internet; telemedicine; mass screening; health behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Masking Description: It is not possible to blind the participants as the intervention is a website. Participants in the intervention arm will need to go through the website and will know its contents while participants in the control arm will not.
  There is no care provider in this study as the intervention is delivered via a website.
  The assignment of intervention or control arm to the participants will be done automatically by the website. After signing the consent form, participants will enter a website which will randomise them to either intervention or control arm. The investigators do not play a role in this.
  The outcome assessment only involves the participants answering a questionnaire themselves. No Outcome Assessor is required to assess any outcome from the participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants who will not be directed to the ScreenMen website
- Intervention group (Experimental): Participants who will be directed to the ScreenMen website
  Interventions: Behavioral: ScreenMen website

INTERVENTIONS:
Behavioral: ScreenMen website — An educational website that aims to improve evidence-based health screening uptake in men
  Arms: Intervention group

SUMMARY:
Health screening is proven to be effective in reducing morbidity, death and healthcare cost. However, the uptake of health screening is low particularly in men. In the earlier phase of this project, a web-based intervention (ScreenMen) to increase health screening uptake in men was developed based on theories, evidence and user needs. It was tested with experts and users for its utility and usability.

In this phase, a randomised controlled trial (RCT) will be conducted to evaluate the effectiveness of ScreenMen in improving health screening knowledge & uptake in men. Healthy men, who have not gone for screening in the past 1 year will be recruited via Facebook to participate in this RCT. The participants will be randomised to receive or not to receive ScreenMen. Knowledge and intention to screen will be measured immediately post-intervention. All participants will be followed up at 1 month and 3 months to measure knowledge, intention and actual uptake of screening.

DETAILED DESCRIPTION:
The uptake of health screening is low in Malaysia, particularly in men. There is a need to increase health screening uptake in men as this will not just save healthcare cost and increase national productivity in the long run but also improve the quality of life of men and their family.

There were many interventions to increase health screening uptake in men which have been identified in the systematic review conducted in the earlier phase of this study. However, there is a lack of ICT-based intervention promoting health screening. The few existing ICT based interventions only focus on screening on a specific disease such as HIV or prostate cancer.(1-3) There was no ICT-based intervention which aimed to increase the uptake of comprehensive health screening.

Studies have shown that ICT-based interventions are effective in improving health behaviour.(4) On top of that, there is a high number of internet accessibility and smartphone ownership in Malaysia, which provides a good platform to promote health screening in men. Thus, ScreenMen, a web-based intervention was developed based on theories, evidence and users' needs. It was tested with experts and users in terms of its utility and usability. (5-7)

To the best of our knowledge, ScreenMen is the first mobile-responsive web-based intervention that promotes comprehensive evidence-based health screening in men. It aims to educate men about screening and empowers them to take charge of their health including undergoing regular health screening. Apart from encouraging health screening, ScreenMen provides advice to men about the recommended health screening they should undergo based on their health risks and educates them to avoid non-evidence-based screening.

Before being launched to the public, a randomised controlled trial (RCT) will be conducted to evaluate the effectiveness of ScreenMen in improving knowledge on screening, intention to screen and the actual uptake of screening. Process evaluation will also be conducted to identify the components that work in improving health screening uptake and resolve any implementation issues of ScreenMen.

ELIGIBILITY:
Inclusion criteria:

* Male
* 18 year old and above
* Own a smart phone

Exclusion criteria:

* Undergone health screening within the past 1 year
* Diagnosed with any of the following diseases (Hypertension, Diabetes, High cholesterol, Colorectal cancer, Lung cancer, Hepatitis B, Hepatitis C, HIV

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants who have undergone health screening | 1 month post-intervention
  A questionnaire will be sent to the participants 1 month after using the intervention (ScreenMen web) to assess whether they have undergone health screening.
  The number of participants who have undergone health screening will be divided over the total number of participants in this study to obtain the proportion and according to study arm.
  Uptake at 1 month Intervention: %= n / N *100%; Control: %= n / N *100%
Number of participants who have undergone health screening | 3 months post-intervention
  Participants who reported that they have not undergone health screening during the 1-month follow up will be followed up at 3-month. They will be asked whether they have undergone health screening up to this stage.
  The number of participants who have undergone health screening (including those from 1-month follow up) will be divided over the total number of participants in this study to obtain the proportion and according to study arm.
  Uptake at 3 month (including those reported yes in 1-month follow up) Intervention: %= n / N *100%; Control: %= n / N *100%

SECONDARY OUTCOMES:
Change in intention (months) to undergo health screening | Immediately post-intervention
  Immediately after using the ScreenMen web, participants will be asked when do they intend to undergo health screening. They will be asked in terms of 'in the next __ month(s)'.
  The same question has been asked pre-intervention. The change in the 'month(s)' will be calculated. This will be averaged and compared between the intervention and control group.
  Change in intention to screen (months) immediately post-intervention = pre-intervention intention to screen (months) - post-intervention intention to screen (months)
  Comparison between the change in intention to screen (months) [immediate] for intervention arm and change in intention to screen (months) [immediate] for control arm will be done.
Change in intention (months) to undergo health screening | 1 month post-intervention
  One month after using the ScreenMen web, participants will be followed up and asked if they have undergone health screening. If not, they will be asked when do they intend to undergo health screening. They will be asked in terms of 'in the next __ month(s)'.
  Change in intention to screen will be calculated based on their immediate intention to screen after intervention
  Comparison between the change in intention to screen (months) [1-month] for intervention arm and change in intention to screen (months) [1-month] for control arm will be done.
  The aim of this is to evaluate the long-term effect of the intervention, whether it is sustained or diminished.
Change in intention (months) to undergo health screening | 3 months post-intervention
  Participants who have not undergone screening will be followed up again at 3-month and asked if they have undergone health screening. If not, they will be asked when do they intend to undergo health screening. They will be asked in terms of 'in the next __ month(s)'.
  Change in intention to screen will be calculated based on their immediate intention to screen after intervention
  Comparison between the change in intention to screen (months) [3-month] for intervention arm and change in intention to screen (months) [3-month] for control arm will be done.
  The aim of this is to evaluate the long-term effect of the intervention, whether it is sustained or diminished.
Change in knowledge on health screening | Immediately post-intervention
  Immediately after using the ScreenMen web, participants will be asked to answer a validated questionnaire on health screening. The score will be calculated by calculating the number of correctly answered questions over the total number of questions. Knowledge Score (post-intervention - immediate) = n/N
  The participants have filled the same questionnaire pre-intervention. Change of knowledge score will be calculated as shown below:
  Change in Knowledge Score = Knowledge Score (post-intervention - immediate) - Knowledge Score (pre-intervention)
  The Change in Knowledge Score will be compared between intervention and control group.
Change in knowledge on health screening | 1 month post-intervention
  One month after using the ScreenMen web, participants will be followed up and asked to fill up the same health screening questionnaire. The score will be calculated by calculating the number of correctly answered questions over the total number of questions. Knowledge Score (post-intervention - immediate) = n/N
  Change of knowledge score from immediate to 1 month post-intervention will be calculated as shown below:
  Change in Knowledge Score = Knowledge Score (1 month post-intervention) - Knowledge Score (immediately post-intervention)
  The Change in Knowledge Score from immediate to 1 month post-intervention will be compared between intervention and control group.
  The aim of this is to evaluate the long-term effect of the intervention, whether the participants' knowledge on health screening is sustained or diminished.
Change in knowledge on health screening | 3 months post-intervention
  Three months after using the ScreenMen web, participants will be followed up and asked to fill up the same health screening questionnaire. The score will be calculated by calculating the number of correctly answered questions over the total number of questions. Knowledge Score (post-intervention - immediate) = n/N
  Change of knowledge score from immediate to 3 months post-intervention will be calculated as shown below:
  Change in Knowledge Score = Knowledge Score (3 months post-intervention) - Knowledge Score (immediately post-intervention)
  The Change in Knowledge Score from immediate to 1 months post-intervention will be compared between intervention and control group.
  The aim of this is to evaluate the long-term effect of the intervention, whether the participants' knowledge on health screening is sustained or diminished.

CONTACTS AND LOCATIONS:
Overall Officials: Chirk Jenn Ng, MMed,PhD, Principal Investigator — University of Malaya
Locations (1):
- University of Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bauermeister JA, Pingel ES, Jadwin-Cakmak L, Harper GW, Horvath K, Weiss G, Dittus P. Acceptability and preliminary efficacy of a tailored online HIV/STI testing intervention for young men who have sex with men: the Get Connected! program. AIDS Behav. 2015 Oct;19(10):1860-74. doi: 10.1007/s10461-015-1009-y. PMID 25638038
- [Background] Evans R, Joseph-Williams N, Edwards A, Newcombe RG, Wright P, Kinnersley P, Griffiths J, Jones M, Williams J, Grol R, Elwyn G. Supporting informed decision making for prostate specific antigen (PSA) testing on the web: an online randomized controlled trial. J Med Internet Res. 2010 Aug 6;12(3):e27. doi: 10.2196/jmir.1305. PMID 20693148
- [Background] Hirshfield S, Chiasson MA, Joseph H, Scheinmann R, Johnson WD, Remien RH, Shaw FS, Emmons R, Yu G, Margolis AD. An online randomized controlled trial evaluating HIV prevention digital media interventions for men who have sex with men. PLoS One. 2012;7(10):e46252. doi: 10.1371/journal.pone.0046252. Epub 2012 Oct 2. PMID 23071551
- [Background] Wantland DJ, Portillo CJ, Holzemer WL, Slaughter R, McGhee EM. The effectiveness of Web-based vs. non-Web-based interventions: a meta-analysis of behavioral change outcomes. J Med Internet Res. 2004 Nov 10;6(4):e40. doi: 10.2196/jmir.6.4.e40. PMID 15631964
- [Background] Schnall R, Rojas M, Bakken S, Brown W, Carballo-Dieguez A, Carry M, Gelaude D, Mosley JP, Travers J. A user-centered model for designing consumer mobile health (mHealth) applications (apps). J Biomed Inform. 2016 Apr;60:243-51. doi: 10.1016/j.jbi.2016.02.002. Epub 2016 Feb 20. PMID 26903153
- [Background] Uhler LM, Perez Figueroa RE, Dickson M, McCullagh L, Kushniruk A, Monkman H, Witteman HO, Hajizadeh N. InformedTogether: Usability Evaluation of a Web-Based Decision Aid to Facilitate Shared Advance Care Planning for Severe Chronic Obstructive Pulmonary Disease. JMIR Hum Factors. 2015 Feb 25;2(1):e2. doi: 10.2196/humanfactors.3842. PMID 27025896
- [Background] Verkuyl M, Atack L, Mastrilli P, Romaniuk D. Virtual gaming to develop students' pediatric nursing skills: A usability test. Nurse Educ Today. 2016 Nov;46:81-85. doi: 10.1016/j.nedt.2016.08.024. Epub 2016 Aug 25. PMID 27614548
- [Background] Young SD, Cumberland WG, Lee SJ, Jaganath D, Szekeres G, Coates T. Social networking technologies as an emerging tool for HIV prevention: a cluster randomized trial. Ann Intern Med. 2013 Sep 3;159(5):318-24. doi: 10.7326/0003-4819-159-5-201309030-00005. PMID 24026317